CLINICAL TRIAL: NCT05247970
Title: A Phase 1 Randomized, Double-blind, Single and Multiple-dose Study to Assess the Safety, Tolerability, Pharmacokinetics, Food Effect, and Drug-Drug Interactions of S-309309 in Healthy and Obese Adult Study Participants
Brief Title: A Study to Assess S-309309 in Healthy and Obese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018N1111
Record Dates: First submitted 2022-02-08; First posted 2022-02-21 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: S-309309 (Experimental): Participants will receive S-309309 at specific timepoints in a fasted state.
  Interventions: Drug: S-309309
- Part 2: S-309309 and Midazolam (Experimental): Participants will receive S-309309 and Midazolam at specific timepoints fed state.
  Interventions: Drug: S-309309; Drug: Midazolam
- Part 1 and 2: Placebo (Placebo Comparator): Participants will receive a matching placebo to S-309309 at specific timepoints in either a fed or fasted state.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-309309 — Capsule administered orally
  Arms: Part 1: S-309309; Part 2: S-309309 and Midazolam
Drug: Midazolam — Syrup administered orally
  Arms: Part 2: S-309309 and Midazolam
Drug: Placebo — Matching capsule to S-309309 administered orally
  Arms: Part 1 and 2: Placebo

SUMMARY:
The primary aim of the study is to assess the safety and tolerability of S-309309 after oral administration in healthy adult or obese but otherwise healthy adult participants. The secondary aim of the study is to assess the pharmacokinetics of S-309309 and the effects on ECG parameters after oral administration in healthy or obese but otherwise healthy participants.

DETAILED DESCRIPTION:
This study will consist of 2 Parts. Part 1 will include healthy participants who will be assigned to a dose group. Participants will then be randomized to receive a single oral administration of S-309309 or placebo in a fasted state. Administration will be initiated in the lowest dose group, and administration in the next dose group will not occur until a review of safety and tolerability has been completed for the preceding group.

Part 2 will include 2 groups. Healthy participants and obese but otherwise healthy participants will receive multiple oral administrations of S-309309 or placebo in a fed state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by medical evaluation including medical history, physical examination, clinical laboratory tests, vital sign measurements, and 12-lead ECG at the Screening Visit and upon admission to the clinical research unit (CRU).
* Body weight ≥50 kilograms (kg), and body mass index (BMI) within the range ≥18.5 to <30.0 kilogram/meter square (kg/m^2) for all groups except Group G-2. For Group G-2, BMI ≥ 30 to < 40 kg/m2 at the Screening Visit.

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* Breast cancer within the past 10 years.
* Unable to swallow capsules.
* Chronic history of or current liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Part 1 and 2: Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to Day 28

SECONDARY OUTCOMES:
Part 1: Maximum Plasma Concentration (Cmax) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Time to Maximum Plasma Concentration (Tmax) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Area Under the Plasma Concentration-Time Curve (AUC) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Terminal Elimination Half-Life (t1/2,z) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Terminal Elimination Rate Constant (λz) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Mean Residence Time (MRT) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Apparent Total Clearance (CL/F) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Apparent Volume of Distribution (Vz/F) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Renal Clearance (CLR) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Fraction of Dose Excreted in Urine (Feu) of S-309309 | 0 (predose) up to 144 hours postdose on Day 1 to Day 21
Part 1: Change From Baseline of Electrocardiogram (ECG) Parameters: QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF), Pulse Rate (PR) Interval, and Combination of the Q, R, and S Waves (QRS) Duration | Baseline, Day 2, 5, 7 and 16
Part 1: Change From Baseline of ECG Parameter: Heart Rate (HR) | Baseline, Day 2, 3, 4, 5, 6, 7 and 16
Part 1: Placebo-Corrected Change From Baseline of ECG Parameters: QTcF, PR Interval, and QRS Duration | Baseline, Day 2, 5, 7 and 16
Part 1: Placebo-Corrected Change From Baseline of ECG Parameter: HR | Baseline, Day 2, 3, 4, 5, 6, 7 and 16
Part 1: Number of Participants With Categorical Outlier Values for HR, QTcF, PR, and QRS | Baseline up to Day 16
Part 1: Number of Participants With Treatment-Emergent Changes for T-wave Morphology and Presence of U-wave | Baseline up to Day 16
Part 2: Cmax of S-309309 and Midazolam | 0 (predose) up to 24 hours postdose on Day -2 to Day 16
Part 2: Tmax of S-309309 and Midazolam | 0 (predose) up to 24 hours postdose on Day -2 to Day 16
Part 2: AUC of S-309309 and Midazolam | 0 (predose) up to 24 hours postdose on Day -2 to Day 16
Part 2: t1/2,z of S-309309 and Midazolam | 0 (predose) up to 24 hours postdose on Day -2 to Day 16
Part 2: λz of S-309309 and Midazolam | 0 (predose) up to 24 hours postdose on Day -2 to Day 16
Part 2: CL/F of S-309309 and Midazolam | 0 (predose) up to 24 hours postdose on Day -2 to Day 16
Part 2: Vz/F of S-309309 and Midazolam | 0 (predose) up to 24 hours postdose on Day -2 to Day 16
Part 2: MRT of Midazolam | 0 (predose) up to 24 hours postdose on Day -2 to Day 16
Part 2: Number of Participants with TEAEs After Coadministration with Midazolam | Up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Early Phase Services, LLC, San Antonio, Texas, United States

REFERENCES:
- [Derived] Ishibashi T, Tanioka H, Ikehara T, Kezbor S, Sonoyama T. Safety, Tolerability, and Pharmacokinetics of a Novel Anti-obesity Agent, S-309309, in Healthy Adults with or Without Obesity. Clin Drug Investig. 2025 Feb;45(2):85-99. doi: 10.1007/s40261-024-01418-3. Epub 2025 Jan 20. PMID 39832041